CLINICAL TRIAL: NCT04493086
Title: Effect of FFRCT-angio in Functional Diagnosis of Coronary Artery Stenosis: a Prospective, Multicenter Clinical Study
Brief Title: Effect of FFRCT-angio in Functional Diagnosis of Coronary Artery Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: FFR
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FFRCT-angio — According to invasive coronary angiography (CAG) images, image databases of critical lesions, diffuse lesions, left main trunk lesions, ostium lesions and bifurcation lesions were established. In order to ensure that the position of the pressure guide wire sensor is consistent with that of FFRCT-angio, a professional with unknown FFR results is used to mark the position of the pressure wire sensor on the CAG image. The clinical information and characteristics of coronary artery lesions were collected, and the baseline data of patients were completed. The accuracy and diagnostic performance of FFRCT-angio in the diagnosis of functional stenosis (FFR < 0.8) were evaluated with FFR value measured by pressure guide wire as reference standard.

SUMMARY:
Coronary CT angiography (CTA) or invasive coronary angiography (CAG) is usually performed to evaluate the severity of coronary stenosis depending on the probability of CAD. However, the stenosis severity is not closely corresponding with the hemodynamic significance in coronary arteries.

As a result, fractional flow reserve (FFR) with pressure wire measurement was introduced to functionally assess the coronary stenosis. FFR is defined as the ratio of maximum blood flow distal to a stenotic lesion under hyperemia state to normal maximum flow in the same vessel. The cutoff value of FFR to detect significant ischemia is set to be 0.80, indicating that PCI should be considered if FFR≤0.80. However, FFR does have some limitations, such as risks of pressure wire injury, extra time and cost, and side effects of hyperemic agents.

To overcome the limitations of FFR, CTA- and CAG-based methods to functionally assess coronary stenosis were proposed, i.e. FFR derived from CTA (FFRCT) and FFR derived from angiography-based quantitative flow ratio (QFR), which can simultaneously evaluate anatomic and hemodynamic significance of stenotic lesions. A number of studies have demonstrated that FFRCT has high sensitivity and specificity in identifying myocardial ischemia. However, the diagnostic accuracy of FFRCT depends on the image quality of coronary CTA, and it is relatively low in lesions with severe calcification and/or tortuosity. Besides, the methodology of FFRCT relies on computational fluid dynamics, which is complicated and time consuming. As for QFR, it is a novel method for deriving FFR based on 3-dimensional quantitative coronary angiography (3D-QCA) and contrast frame counting during CAG. Recent studies have shown that QFR has good diagnostic performance in evaluating the functional significance of coronary stenosis. The accuracy of QFR is also highly associated with anatomic information, thereby its diagnostic accuracy may be decreased in diffuse, tandem, thrombus-containing, calcified, or torturous lesions, and it is not suitable for prior infarction-related or collateral donor arteries as well. Given the above issues concerning FFRCT and QFR, we proposed a novel approach that integrates coronary CTA and CAG images to calculate FFR (FFRCT-angio) using artificial intelligence. The present study was undertaken to test the diagnostic accuracy of FFRCT-angio in patients with SCAD.

DETAILED DESCRIPTION:
Cardiovascular disease remains the leading cause of death worldwide, and stable coronary artery disease (SCAD) accounts for the greatest proportion of cardiovascular disease. In the past decades, percutaneous coronary intervention (PCI) has become one of the most common treatments for SCAD, and therefore assessing the hemodynamic significance of coronary stenosis is important for physicians to make the optimal treating strategy. Coronary CT angiography (CTA) or invasive coronary angiography (CAG) is usually performed to evaluate the severity of coronary stenosis depending on the probability of CAD. However, the stenosis severity is not closely corresponding with the hemodynamic significance in coronary arteries.

As a result, fractional flow reserve (FFR) with pressure wire measurement was introduced to functionally assess the coronary stenosis. FFR is defined as the ratio of maximum blood flow distal to a stenotic lesion under hyperemia state to normal maximum flow in the same vessel. The cutoff value of FFR to detect significant ischemia is set to be 0.80, indicating that PCI should be considered if FFR≤0.80. FAME (Fractional Flow Reserve versus Angiography for Multivessel Evaluation) study confirmed that FFR guided PCI was superior to angiography guided PCI in reducing major adverse cardiovascular events (MACE) in patients with multivessel disease. In the subsequent FAME 2 study, FFR guided PCI plus the optimal medical treatment (OMT), as compared with the OMT alone, decreased the composite event rates mainly driven by urgent revascularization in SCAD patients. However, FFR does have some limitations, such as risks of pressure wire injury, extra time and cost, and side effects of hyperemic agents.

To overcome the limitations of FFR, CTA- and CAG-based methods to functionally assess coronary stenosis were proposed, i.e. FFR derived from CTA (FFRCT) and FFR derived from angiography-based quantitative flow ratio (QFR), which can simultaneously evaluate anatomic and hemodynamic significance of stenotic lesions. A number of studies have demonstrated that FFRCT has high sensitivity and specificity in identifying myocardial ischemia. However, the diagnostic accuracy of FFRCT depends on the image quality of coronary CTA, and it is relatively low in lesions with severe calcification and/or tortuosity. Besides, the methodology of FFRCT relies on computational fluid dynamics, which is complicated and time consuming. As for QFR, it is a novel method for deriving FFR based on 3-dimensional quantitative coronary angiography (3D-QCA) and contrast frame counting during CAG. Recent studies have shown that QFR has good diagnostic performance in evaluating the functional significance of coronary stenosis. The accuracy of QFR is also highly associated with anatomic information, thereby its diagnostic accuracy may be decreased in diffuse, tandem, thrombus-containing, calcified, or torturous lesions, and it is not suitable for prior infarction-related or collateral donor arteries as well. Given the above issues concerning FFRCT and QFR, we proposed a novel approach that integrates coronary CTA and CAG images to calculate FFR (FFRCT-angio) using artificial intelligence. The present study was undertaken to test the diagnostic accuracy of FFRCT-angio in patients with SCAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable coronary heart disease undergoing CTA.
* Patients with at least one coronary artery stenosis of 50% - 90% in diameter ≥ 2mm.
* Within 30 days after CTA, CAG and FFR were determined by clinicians according to their condition.

Exclusion Criteria:

* Patients with myocardial infarction within 72 hours.
* Patients with coronary artery thrombosis.
* Patients with a history of allergy to contrast media or adenosine.
* NYHA class III-IV patients.
* Patients with previous CABG, target vessel PCI, pacemaker, ICD.
* Patients with a history of prosthetic valve implantation.
* Patients with myocardial bridges in the target vessels.
* Patients with severe arrhythmia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
By taking FFR value as the standard, evaluating the accuracy of FFRCT-angio in the functional significance of coronary stenosis | 5 days
  By taking FFR value as the standard, evaluating the accuracy of FFRCT-angio in the functional significance of coronary stenosis

SECONDARY OUTCOMES:
By taking FFR value as the standard, evaluating the sensitivity and specificity of FFRCT-angio in the functional significance of coronary stenosis | 5 days
  By taking FFR value as the standard, evaluating the sensitivity and specificity of FFRCT-angio in the functional significance of coronary stenosis

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China